CLINICAL TRIAL: NCT04027439
Title: A Phase II, Randomized Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of Single and Repeat Doses of RPL554 Administered by Dry Powdered Inhaler in Patients With COPD
Brief Title: Study Evaluating 5 Doses of RPL554 and Placebo in COPD Patients Via a Dry Powder Inhaler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RPL554-DP-201
Record Dates: First submitted 2019-03-09; First posted 2019-07-22 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: RPL554 (Active Comparator): Placebo controlled, parallel group single dose. Five of the 6 treatment arms will be double-blind and one will be single-blind
  Interventions: Drug: Part A: RPL554; Drug: Placebos
- Part B: RPL554 (Active Comparator): Double-blind, placebo-controlled, complete block cross-over
  Interventions: Drug: Part B: RPL554; Drug: Placebos

INTERVENTIONS:
Drug: Part A: RPL554 — 1 dose of either 50mcg/100mcg/1500mcg/3000mcg/6000mcg or placebo via dry powder inhaler
  Arms: Part A: RPL554
Drug: Part B: RPL554 — Patients will receive 4 or 5 repeat dose treatments in crossover fashion - doses will be confirmed after Part A
  Arms: Part B: RPL554
Drug: Placebos — Part A: 1 dose of either 50ncg/100ncg/1500ncg/3000ncg/6000ncg or placebo via dry powder inhaler.
  Part B: Patients will receive 4 or 5 repeat dose treatments in crossover fashion - doses will be confirmed after Part A.

SUMMARY:
The purpose of this study is to investigate 5 doses of RPL554 and placebo, administered by dry powder inhaler (DPI), in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The study will consist of two parts. Part A is a parallel group, placebo-controlled single dose study to ascertain the Pharmacokinetics (PK) profile, safety and bronchodilator effect of RPL554 administered via dry powder inhaler (DPI). Five of the 6 treatment arms will be double-blind and one will be single-blind (due to the different number of capsules administered). Part B is a placebo-controlled, complete block cross-over, repeat dose study to assess the bronchodilator effect of repeat doses of RPL554 delivered via a DPI.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
2. For males, not to donate sperm and either be sexually abstinent or use contraception as specified by the protocol. For females, be of non-childbearing potential or use a highly effective form of contraception
3. 12-lead ECG with heart rate between 45 and 90 beats per minute, QTcF ≤450 msec for males, and ≤ 470 msec for females, QRS interval ≤120 msec and no clinically significant abnormality including morphology
4. Capable of complying with all study restrictions and procedures including ability to use the DPI correctly.
5. Body mass index (BMI) between 18 and 35 kg/m2 (inclusive) with a minimum weight of 45 kg.
6. COPD diagnosis for 1 year [prior to screening
7. Ability to perform acceptable and reproducible spirometry.
8. Post-bronchodilator (four puffs of albuterol) spirometry at Screening demonstrating the following:

   * FEV1/Forced Vital Capacity (FVC) ratio of ≤0.70
   * FEV1 ≥40 % and ≤80% of predicted normal
   * ≥150 mL increase from pre-bronchodilator FEV1
9. Clinically stable COPD in the 4 weeks prior to Screening and during the period between Screening and Part A.
10. A chest X-ray showing no abnormalities, which are both clinically significant and unrelated to COPD.
11. Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
12. Current and former smokers with smoking history of ≥10 pack years. 14. Capable of withdrawing from long acting bronchodilators for the duration of the study, and short acting bronchodilators for 8 hours prior to dosing.

Exclusion Criteria:

1. A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
2. COPD exacerbation requiring oral or parenteral steroids, or lower respiratory tract infection requiring antibiotics, within 3 months of Screening or prior to Part A.
3. A history of one or more hospitalizations for COPD or pneumonia within 6 months of Screening or prior to Part A.
4. Intolerance or hypersensitivity to tiotropium, olodaterol, atropine, ipratropium, or RPL554.
5. Evidence of cor pulmonale or clinically significant pulmonary hypertension.
6. Other respiratory disorders
7. Previous lung resection or lung reduction surgery.
8. Use of immunosuppressive therapy, including oral corticosteroids
9. Pulmonary rehabilitation, unless such treatment has been stable from 4 weeks prior to Screening and remains stable during the study.
10. History of, or reason to believe a patient has, drug or alcohol abuse within the past 5 years.
11. Received an experimental drug within 30 days or five half lives, whichever is longer.
12. Patients with uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the Investigator believes are clinically significant.
13. Documented cardiovascular disease, including any history of arrhythmias, angina, recent (<1 year) or suspected myocardial infarction, congestive heart failure, unstable or uncontrolled hypertension, or diagnosis of hypertension within 3 months prior to Screening
14. Use of non-selective oral β-blockers.
15. Major surgery (requiring general anesthesia) within 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
16. A disclosed history or one known to the Investigator, of significant non compliance in previous investigational studies or with prescribed medications.
17. Required use of oxygen therapy, even on an occasional basis.
18. History of malignancy of any organ system within 5 years, with the exception of localized skin cancers (basal or squamous cell).
19. Clinically significant abnormal values for safety laboratory tests (hematology, biochemistry, viral serology or urinalysis) at Screening, as determined by the Investigator. In particular, alanine aminotransferase or aspartate aminotransferase cannot be more than twice the upper limit of normal.
20. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Boscia, MD, Principal Investigator — Vitalink Research
Locations (1):
- VitaLink Research -- Union, Union, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 subjects enrolled for Part A and anticipated to continue into Part B.
Pre-assignment Details: Part A: 37 Patients randomized equally to receive a single dose of RPL554 (0.15, 0.5, 1.5, 3, or 6 mg) or matching placebo via dry powder inhaler (DPI). Patients were to continue to Part B after Part A is complete.
  Part B: 35 Patients continued from Part A and randomly assigned to 1 of 10 treatment sequences in a crossover design (5 x 1-week treatment periods separated by 7-10 day washout). Each sequence included twice daily RPL554 (0.15, 0.5, 1.5, or 3 mg) or matching placebo via DPI.
Groups:
- 0.15 mg/Part A; 0.50 mg/Part A; 1.5 mg/Part A; 3 mg/Part A: Part A: Single dose of RPL554 via DPI (double-blind).
- 6 mg/Part A: Part A: Single dose of RPL554 via DPI (single-blind). Part B: dose not used.
- Placebo/Part A: Part A: Single dose via DPI (double-blind).
- Seq. 1/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 1 = RPL554 .15 mg/1.5 mg/3.0 mg/.50 mg/Placebo.
- Seq. 2/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 2 = RPL554 .15 mg/3.0 mg/Placebo/.50 mg/1.5 mg.
- Seq. 3/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 3 = RPL554 .50 mg/3.0 mg/.15 mg/Placebo/1.5 mg.
- Seq. 4/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 4 = RPL554 .50 mg/.15 mg/1.5 mg/Placebo/3.0 mg.
- Seq. 5/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 5 = RPL554 1.5 mg/.50 mg/Placebo/3.0 mg/.15 mg.
- Seq. 6/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 6 = RPL554 1.5 mg/Placebo/.15 mg/3.0 mg/.50 mg.
- Seq. 7/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 7 = RPL554 3.0 mg/1.5 mg/.50 mg/.15 mg/Placebo.
- Seq. 8/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 8 = RPL554 3.0 mg/Placebo/1.5 mg/.15 mg/.50 mg.
- Seq. 9/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 9 = Placebo/.15 mg/.50 mg/1.5 mg/3.0 mg.
- Seq. 10/Part B: Part B: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over.
  Seq 10 = Placebo/.50 mg/3.0 mg/1.5 mg/.15 mg.
Period: Part A (R, PC, PG) Single Dose
Arm/Group | 0.15 mg/Part A | 0.50 mg/Part A | 1.5 mg/Part A | 3 mg/Part A | 6 mg/Part A | Placebo/Part A | Seq. 1/Part B | Seq. 2/Part B | Seq. 3/Part B | Seq. 4/Part B | Seq. 5/Part B | Seq. 6/Part B | Seq. 7/Part B | Seq. 8/Part B | Seq. 9/Part B | Seq. 10/Part B
Started (Started Part A) | 6 | 6 | 7 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Part A) | 6 | 6 | 7 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (R, PC, CO) Twice Daily for 7 Day
Arm/Group | 0.15 mg/Part A | 0.50 mg/Part A | 1.5 mg/Part A | 3 mg/Part A | 6 mg/Part A | Placebo/Part A | Seq. 1/Part B | Seq. 2/Part B | Seq. 3/Part B | Seq. 4/Part B | Seq. 5/Part B | Seq. 6/Part B | Seq. 7/Part B | Seq. 8/Part B | Seq. 9/Part B | Seq. 10/Part B
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 4 | 3 | 4 | 3 | 3 | 4 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 (1 patient discontinued in part b/period 2 and another in part b/period 3.) | 4 | 3 | 4 | 3 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.15 mg: Single dose of RPL554 via DPI (double-blind)
- 0.50 mg; 1.5 mg; 3 mg: Single dose of RPL554 via DPI (double blind)
- 6 mg: Single dose of RPL554 via DPI (single blind)
- Placebo: Single dose via DPI (double blind)
- Total: Total of all reporting groups
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.15) | 58.3 (3.56) | 63.7 (6.68) | 52.7 (3.88) | 59.3 (7.81) | 60.8 (8.80) | 59.5 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 5 | 2 | 4 | 23
  Male | 2 | 1 | 4 | 1 | 4 | 2 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 0 | 2
  White | 6 | 6 | 5 | 6 | 6 | 6 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 6 | 6 | 6 | 37

OUTCOME MEASURES:

1. Primary Outcome: Part A: RPL554 Plasma Pharmacokinetic Parameter (AUC0-12)
Description: RPL554 Plasma pharmacokinetics AUC0-12 (Area under the Curve) after single dose
Time Frame: Day 1
Population: Pharmacokinetic (PK) Analysis Set in Part A: all randomized patients who had blood sampling performed after the single dose of RPL554 and had evaluable PK parameter data. The PK Analysis Set included the 31 patients who received RPL554 in Part A but not the 6 patients in the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
h*pg/mL | 260 (53.5) | 472 (106.7) | 2210 (62.3) | 4160 (47.2) | 9730 (62.3)

2. Primary Outcome: Part A: RPL554 Plasma Pharmacokinetic Parameter (AUC 0-t)
Description: RPL554 Area under the curve at maximum concentration after a single dose
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
h*pg/mL | 222 (55.5) | 495 (128.2) | 2680 (56.5) | 4920 (44.5) | 11600 (68.3)

3. Primary Outcome: Part A: RPL554 Plasma Pharmacokinetic Parameter (Half-life)
Description: RPL554 Plasma pharmacokinetics Half-life concentration after a single dose
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg
Number analyzed (Participants) | 1 | 5 | 7 | 6 | 6
h | 3.59 | 5.39 (28.7) | 7.48 (43.3) | 6.65 (33.6) | 6.66 (25.4)

4. Primary Outcome: Part B: Change From Baseline in Peak FEV1 (Over 4 Hours)
Description: Change from Baseline FEV1 to Peak FEV1 (over 4 hours) on Day 7
Time Frame: Day 7
Population: All efficacy analyses were carried out using the Full Analysis Set (FAS) in Part B: all randomized patients with sufficient data (pre-dose and at least 1 post-dose assessment of spirometry) collected after intake of study medication to compute the PD parameters (FEV1, FRC measurements) on at least 2 treatment periods in Part B. The FAS comprised: RPL554 0.15 mg (N=34); RPL554 0.5 mg (N=33); RPL554 1.5 mg (N=32); RPL554 3 mg (N=33); Placebo (N=32).
Measure: Mean (Standard Deviation); unit: L
Groups:
- 0.15 mg; 0.50 mg; 1.5 mg; 3 mg: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over
- Placebo: 7 day, twice daily dose of placebo via DPI (double-blind) complete block, cross-over
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 31 | 32 | 32
L | 0.220 (0.1593) | 0.293 (0.2411) | 0.298 (0.2355) | 0.378 (0.2182) | 0.118 (0.1437)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.186, 95% CI 2-sided [1.138 to 1.235]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.134, 95% CI 2-sided [1.088 to 1.181]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.134, 95% CI 2-sided [1.089 to 1.181]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.0001, ANCOVA; Contrast Ratio = 1.084, 95% CI 2-sided [1.041 to 1.128]

5. Secondary Outcome: Part A: Change From Baseline in Average FEV1 (Over 4 Hours)
Description: Change from Baseline FEV1 to Average FEV1 (over 4 hours) After Single Dose
Time Frame: Day 1
Population: Full Analysis Set (FAS) in Part A: all randomized patients with sufficient data collected after intake of study medication to compute the PD parameters (FEV1 measurements pre dose and at least 1 post-baseline). All 37 patients randomized into Part A were included in the FAS.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6
L | 0.109 (0.0380) | 0.213 (0.1226) | 0.326 (0.249) | 0.337 (0.1831) | 0.334 (0.1170) | 0.040 (0.0517)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p = 0.0004, ANCOVA; Contrast Ratio = 1.228, 95% CI 2-sided [1.105 to 1.365]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0004, ANCOVA; Contrast Ratio = 1.228, 95% CI 2-sided [1.104 to 1.365]
Statistical Analysis 3: Comparison: 1.5 mg vs Placebo; Test type: Other; p = 0.0012, ANCOVA; Contrast Ratio = 1.196, 95% CI 2-sided [1.080 to 1.326]
Statistical Analysis 4: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.0348, ANCOVA; Contrast Ratio = 1.121, 95% CI 2-sided [1.009 to 1.246]
Statistical Analysis 5: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.3106, ANCOVA; Contrast Ratio = 1.055, 95% CI 2-sided [0.949 to 1.172]

6. Secondary Outcome: Part A: Change From Baseline in Average FEV1 (Over 12 Hours)
Description: Change from Baseline FEV1 to Average FEV1 (over 12 hours) After Single Dose
Time Frame: Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6
L | 0.045 (0.0384) | 0.113 (0.1703) | 0.214 (0.2172) | 0.243 (0.2715) | 0.176 (0.0481) | -0.011 (0.0749)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p = 0.0208, ANCOVA; Contrast Ratio = 1.154, 95% CI 2-sided [1.024 to 1.301]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0041, ANCOVA; Contrast Ratio = 1.200, 95% CI 2-sided [1.064 to 1.353]
Statistical Analysis 3: Comparison: 1.5 mg vs Placebo; Test type: Other; p = 0.0108, ANCOVA; Contrast Ratio = 1.167, 95% CI 2-sided [1.039 to 1.311]
Statistical Analysis 4: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.1641, ANCOVA; Contrast Ratio = 1.087, 95% CI 2-sided [0.965 to 1.225]

7. Secondary Outcome: Part A: Change From Baseline in Peak FEV1 (Over 4 Hours)
Description: Change from Baseline FEV1 to Peak FEV1 (over 4 hours) After Single Dose
Time Frame: Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6
L | 0.203 (0.0646) | 0.298 (0.1280) | 0.429 (0.2504) | 0.468 (0.2135) | 0.452 (0.1382) | 0.135 (0.0922)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p = 0.0005, ANCOVA; Contrast Ratio = 1.229, 95% CI 2-sided [1.102 to 1.369]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0005, ANCOVA; Contrast Ratio = 1.231, 95% CI 2-sided [1.104 to 1.372]
Statistical Analysis 3: Comparison: 1.5 mg vs Placebo; Test type: Other; p = 0.0022, ANCOVA; Contrast Ratio = 1.188, 95% CI 2-sided [1.070 to 1.320]
Statistical Analysis 4: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.0658, ANCOVA; Contrast Ratio = 1.106, 95% CI 2-sided [0.993 to 1.233]

8. Secondary Outcome: Part A: Safety and Tolerability / Hematology Safety Assessments
Description: number of patients with treatment-emergent hematology abnormal laboratory assessments
Time Frame: Day 1
Reporting Status: Not Posted

9. Secondary Outcome: Part A: Safety and Tolerability / Blood Chemistry Safety Assessments
Description: number of patients with treatment-emergent blood chemistry abnormal laboratory assessments
Time Frame: Day 1
Reporting Status: Not Posted

10. Secondary Outcome: Part A: Safety and Tolerability / Urinalysis Safety Assessments
Description: number of patients with treatment-emergent urinalysis abnormal laboratory assessments
Time Frame: Day 1
Reporting Status: Not Posted

11. Secondary Outcome: Part A: Safety and Tolerability / Supine Vital Signs - Pulse Rate
Description: Change from Baseline Pulse Rate to Peak Pulse Rate (over 4 hours) After Single Dose
Time Frame: Day 1
Reporting Status: Not Posted

12. Secondary Outcome: Part A: Safety and Tolerability / Supine Vital Signs - Blood Pressure
Description: number of patients with treatment-emergent abnormal vital signs (blood pressure in mm Hg) (An increase from baseline of >=20 in systolic bp)
Time Frame: Day 1
Reporting Status: Not Posted

13. Secondary Outcome: Part A: Safety and Tolerability / ECG - QTcF
Description: number of patients with treatment-emergent abnormal ECG parameters, QTcF in msec
Time Frame: Day 1
Reporting Status: Not Posted

14. Secondary Outcome: Part A: Safety and Tolerability / ECG - Heart Rate
Description: number of patients with treatment-emergent clinically significant abnormal ECG parameters, heart rate in bpm
Time Frame: Day 1
Reporting Status: Not Posted

15. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 4 Hrs)
Description: Change from baseline in average FEV1 (over 4 hours) on Day 7
Time Frame: Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 31 | 32 | 32
L | 0.100 (0.1430) | 0.176 (0.2253) | 0.184 (0.2176) | 0.244 (0.1953) | 0.017 (0.1526)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.183, 95% CI 2-sided [1.134 to 1.234]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.140, 95% CI 2-sided [1.092 to 1.190]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.131, 95% CI 2-sided [1.084 to 1.180]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.0004, ANCOVA; Contrast Ratio = 1.080, 95% CI 2-sided [1.036 to 1.126]

16. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 12 Hours)
Description: Change from baseline FEV1 in average FEV1 (over 12 hours) on Day 7
Time Frame: Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 31 | 32 | 32
L | 0.052 (0.1759) | 0.106 (0.2125) | 0.096 (0.1796) | 0.163 (0.1679) | 0.016 (0.1455)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.123, 95% CI 2-sided [1.078 to 1.169]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p = 0.0004, ANCOVA; Contrast Ratio = 1.078, 95% CI 2-sided [1.035 to 1.122]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.0002, ANCOVA; Contrast Ratio = 1.081, 95% CI 2-sided [1.039 to 1.125]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.0437, ANCOVA; Contrast Ratio = 1.041, 95% CI 2-sided [1.001 to 1.083]

17. Secondary Outcome: Part B: Change From Baseline in Trough FEV1
Description: Change from Baseline FEV1 to Morning Trough FEV1 on Day 7
Time Frame: Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 32 | 31 | 32 | 32
L | -0.036 (0.1332) | 0.031 (0.1821) | 0.020 (0.1838) | 0.030 (0.1539) | -0.067 (0.1577)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0006, ANCOVA; Contrast Ratio = 1.087, 95% CI 2-sided [1.038 to 1.139]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p = 0.0010, ANCOVA; Contrast Ratio = 1.083, 95% CI 2-sided [1.034 to 1.135]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.0002, ANCOVA; Contrast Ratio = 1.096, 95% CI 2-sided [1.047 to 1.149]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.0971, ANCOVA; Contrast Ratio = 1.039, 95% CI 2-sided [0.993 to 1.088]

18. Secondary Outcome: Part B: Change From Baseline in Peak FEV1 (Over 4 Hours)
Description: Change from baseline FEV1 in peak FEV1 (over 4 hours) after first dose
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 32 | 33 | 32
L | 0.310 (0.1382) | 0.332 (0.2181) | 0.401 (0.1705) | 0.404 (0.1867) | 0.188 (0.1267)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.145, 95% CI 2-sided [1.106 to 1.185]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.148, 95% CI 2-sided [1.109 to 1.189]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.099, 95% CI 2-sided [1.062 to 1.137]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.088, 95% CI 2-sided [1.052 to 1.126]

19. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 4 Hours)
Description: Change from baseline FEV1 in average FEV1 (over 4 hours) on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 32 | 33 | 32
L | 0.201 (0.1180) | 0.227 (0.2026) | 0.268 (0.1518) | 0.285 (0.1597) | 0.079 (0.1081)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.150, 95% CI 2-sided [1.113 to 1.189]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.146, 95% CI 2-sided [1.109 to 1.185]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.107, 95% CI 2-sided [1.071 to 1.144]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.094, 95% CI 2-sided [1.059 to 1.130]

20. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 12 Hours)
Description: Change from baseline FEV1 in average FEV1 (over 12 hours) on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 32 | 33 | 32
L | 0.101 (0.1314) | 0.139 (0.1921) | 0.135 (0.1655) | 0.182 (0.1536) | 0.044 (0.1073)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.103, 95% CI 2-sided [1.066 to 1.141]
Statistical Analysis 2: Comparison: 1.5 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; Contrast Ratio = 1.078, 95% CI 2-sided [1.042 to 1.116]
Statistical Analysis 3: Comparison: 0.50 mg vs Placebo; Test type: Other; p = 0.0002, ANCOVA; Contrast Ratio = 1.067, 95% CI 2-sided [1.032 to 1.104]
Statistical Analysis 4: Comparison: 0.15 mg vs Placebo; Test type: Other; p = 0.0066, ANCOVA; Contrast Ratio = 1.048, 95% CI 2-sided [1.013 to 1.084]

21. Secondary Outcome: Part B: RPL554 Plasma Pharmacokinetic Parameter (Onset of Action)
Description: Determination of onset of action (>10% increase in FEV1 from pre- to post-first dose, censored at 120 minutes) on Day 1
Time Frame: Day 1
Population: Pharmacokinetic (PK) Analysis Set in Part B: all randomized patients who had blood sampling performed after at least 1 dose of RPL554 in Part B and with data sufficient to calculate PK parameters. The PK analysis set comprised: RPL554 0.15 mg (N=34); RPL554 0.5 mg (N=33); RPL554 1.5 mg (N=32); RPL554 3 mg (N=33); Placebo (N=32).
Measure: Median (Full Range); unit: mins
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg
Number analyzed (Participants) | 29 | 27 | 30 | 31
mins | 13.0 [3 to 120] | 15 [3 to 120] | 15 [4 to 125] | 13 [4 to 120]

22. Secondary Outcome: Part B: Safety and Tolerability / Hematology Safety Assessments
Description: number of patients with treatment-emergent hematology abnormal laboratory assessments (changes from normal at baseline to low or high on Day 7 or at the end of study in >3 patients in each treatment group).
Time Frame: Day 7
Reporting Status: Not Posted

23. Secondary Outcome: Part B: Safety and Tolerability / Blood Chemistry Safety Assessments
Description: number of patients with treatment-emergent blood chemistry abnormal laboratory assessments (changes from normal at baseline to low or high on Day 7 in each treatment group).
Time Frame: Day 7
Reporting Status: Not Posted

24. Secondary Outcome: Part B: Safety and Tolerability / Urinalysis Safety Assessments
Description: number of patients with treatment-emergent urinalysis abnormal laboratory assessments
Time Frame: Day 7
Reporting Status: Not Posted

25. Secondary Outcome: Part B: Safety and Tolerability / ECG - QTcF
Description: number of patients with treatment-emergent clinically significant abnormal ECG parameters, QTcF in msec
Time Frame: Day 7
Reporting Status: Not Posted

26. Secondary Outcome: Part B: Safety and Tolerability / ECG - Heart Rate
Description: number of patients with treatment-emergent abnormal ECG parameters, heart rate in bpm
Time Frame: Day 7
Reporting Status: Not Posted

27. Secondary Outcome: Part B: Safety and Tolerability / Supine Vital Signs - Pulse Rate
Description: number of patients with treatment-emergent abnormal vital signs (pulse rate in bpm) An increase from baseline of >=20
Time Frame: Day 7
Reporting Status: Not Posted

28. Secondary Outcome: Part B: Safety and Tolerability / Supine Vital Signs - Blood Pressure
Description: number of patients with treatment-emergent abnormal vital signs (systolic blood pressure in mm Hg) (An increase from baseline of >=20)
Time Frame: Day 7
Reporting Status: Not Posted

29. Secondary Outcome: Part B: Change From Baseline in Peak Pulse Rate (Day 1)
Description: Change from baseline in peak pulse after first dose on Day 1
Time Frame: Day 1
Reporting Status: Not Posted

30. Secondary Outcome: Part B: Change From Baseline in Peak Pulse Rate (Day 7)
Description: Change from baseline in peak pulse after morning dosing on Day 7
Time Frame: Day 7
Reporting Status: Not Posted

31. Secondary Outcome: Part B: RPL554 Plasma Pharmacokinetic Parameter (Tmax)
Description: RPL554 steady-state PK (tmax) after morning dose on Day 7
Time Frame: Day 7
Population: as for outcome 21
Measure: Median (Full Range); unit: h
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg
Number analyzed (Participants) | 33 | 31 | 30 | 31
h | 1.000 [0.417 to 2.000] | 1.000 [0.000 to 3.917] | 1.000 [0.000 to 2.000] | 1.000 [0.000 to 2.000]

32. Secondary Outcome: Part B: RPL554 Plasma Pharmacokinetic Parameter (Cmax)
Description: RPL554 steady-state PK (Cmax and accumulation ratio) after morning dose on Day 7
Time Frame: Day 7
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg
Number analyzed (Participants) | 33 | 31 | 30 | 31
pg/mL | 68.7 (41.6) | 237 (47.4) | 591 (71.1) | 1240 (41.4)

33. Secondary Outcome: Part B: RPL554 Plasma Pharmacokinetic Parameter (AUC0-12h)
Description: RPL554 steady-state PK (AUC0-12h and accumulation ratio) after morning dose on Day 7
Time Frame: Day 7
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | 0.15 mg | 0.50 mg | 1.5 mg | 3 mg
Number analyzed (Participants) | 33 | 31 | 30 | 31
h*pg/mL | 263 (56.2) | 1240 (52.3) | 3070 (73.6) | 6460 (49.9)

ADVERSE EVENTS:
Time Frame: Part A: 24 hours. Part B: Approximately 70 days
Groups:
- Part A: 0.15 mg: Single dose of RPL554 via DPI (double-blind)
- Part A: 0.50 mg; Part A: 1.5 mg; Part A: 3 mg: Single dose of RPL554 via DPI (double blind)
- Part A: 6 mg: Single dose of RPL554 via DPI (single blind)
- Part A: Placebo: Single dose of placebo via DPI (double blind)
- Part B: 0.15 mg; Part B: 0.50 mg; Part B: 1.5 mg; Part B: 3 mg: 7 day, twice daily dose of RPL554 via DPI (double-blind) complete block, cross-over
- Part B: Placebo: 7 day, twice daily dose of placebo via DPI (double-blind) complete block, cross-over
Arm/Group | Part A: 0.15 mg | Part A: 0.50 mg | Part A: 1.5 mg | Part A: 3 mg | Part A: 6 mg | Part A: Placebo | Part B: 0.15 mg | Part B: 0.50 mg | Part B: 1.5 mg | Part B: 3 mg | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/35 | 0/33 | 0/32 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/35 | 0/33 | 0/32 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/7 | 0/6 | 0/6 | 0/6 | 3/35 | 9/33 | 4/32 | 4/33 | 5/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 0.15 mg (N=6) | Part A: 0.50 mg (N=6) | Part A: 1.5 mg (N=7) | Part A: 3 mg (N=6) | Part A: 6 mg (N=6) | Part A: Placebo (N=6) | Part B: 0.15 mg (N=35) | Part B: 0.50 mg (N=33) | Part B: 1.5 mg (N=32) | Part B: 3 mg (N=33) | Part B: Placebo (N=32)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT04027439/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04027439/SAP_001.pdf